CLINICAL TRIAL: NCT04756440
Title: The Effect of Music Therapy and Planned Education Program on Roma Women's Awareness and Health Beliefs Regarding Cervical Cancer and Screening
Brief Title: The Effect of the Program on the Awareness of Roma Women on Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Ilknur Aydin Avci, Head of Nursing Department, Ondokuz Mayıs University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: B.30.2.ODM.0.20.08/616-704
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Cervical Cancer
Keywords: Roma women; music therapy; early screening; cancer; awareness; health belief model
MeSH Terms: conditions — Uterine Cervical Neoplasms; Neoplasms | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled experimental design
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Intervention Group (Experimental): Firstly, Pre-tests were applied to the women in the experimental group. The 4-week training program created by taking into account the cultural characteristics of the Roma; It includes the Anatomy of Female Reproductive Organs, Anatomy of the Cervix, Cancer, Cervical Cancer, Early diagnosis and its importance, Pap smear test, HPV-DNA test, Cancer Early Diagnosis, Screening and Education Center. Afterwards, music therapy will be applied to the women in the experimental group with the song written and composed by the researchers who emphasized the importance of early diagnosis. At the end of the program, a focus group discussion will be held with the participants in the experimental group regarding their educational experiences, learning experiences for cervical cancer and screening, and program outcomes. Final tests will be made 3 months after the training ends.
  Interventions: Behavioral: Education Program and Music Therapy
- No Intervention: Control Group (No Intervention): First, pre-tests will be applied to the women in the control group. Women in this group will not be intervened and post-tests will be made 3 months after the pre-test.

INTERVENTIONS:
Behavioral: Education Program and Music Therapy — After the intervention, it is expected that their awareness of Romana cervical cancer will increase, their perception of obstacle towards screening tests will decrease and they will be tested.
  Arms: Experimental: Intervention Group

SUMMARY:
This study, which is designed according to the experimental model with randomized pre-test and post-test control group, will be carried out with Roman women who apply to Yavuz Selim Family Health Center in Samsun province, Canik district, where Roma citizens are densely registered.The population of the study consists of Roma women aged 30-65 who are registered to Yavuz Selim Family Health Center in Canik district of Samsun province. The working group will be composed of 80 Roma women who meet the selection criteria. The turkey in cervical cancer screening taking rate is 50% and 17% to 5% error when Roman population was identified as sample size 62 with power 80%.Since the study will consist of experiment and control groups, each group will be determined as 31 people, and 9 backups will be taken, considering that there may be losses. As a result, the research will be conducted as 40 people in the experimental group and 40 people in the control group.A personal questionnaire prepared by the researcher in line with the literature, Cervical Cancer and Pap Smear Test Health Belief Model Scale will be applied to the Roma women who apply to Yavuz Selim Family Health Center and who have accepted to participate in the study by explaining the purpose of the research and those who accept to participate in the study. Roma women who are pre-tested will be randomly assigned to the sample pool to be divided into experimental and control groups. Roman women will be divided into experimental and control groups by Simple Random Method.A 4-week training program will be applied to the experimental group. Afterwards, 2 weeks of training will be done through music. At the end of the training, a focus group discussion will be held with the participants in the experimental group regarding their educational experiences, learning experiences for cervical cancer and screening and program outcomes.A personal questionnaire, Cervical Cancer and Pap Smear Test Health Belief Model Scale will be applied to the experimental and control groups as a final test.

DETAILED DESCRIPTION:
In this study, it is aimed to present an innovative approach in ensuring the participation of Roma women in cervical cancer screenings. For this purpose, music therapy and planned education program will be implemented in order to influence the health beliefs of Roma women.Study design ans setting The research was conducted in a randomized controlled double-blind pretest-posttest controlor the control group. The randomized clinical trial was based on the guidelines proposed by the Consolidated standard of Reporting Trials- CONSORT 2010. The data of the study will be collected in Samsun / Canik District Yavuz Selim Family Health Center between January and June 2021.

A personal questionnaire prepared by the researcher in line with the literature, Cervical Cancer and Pap Smear Test Health Belief Model Scale will be applied to the Roma women who apply to Yavuz Selim Family Health Center and who have accepted to participate in the study by explaining the purpose of the research and those who accept to participate in the study. Pre-tests will be done to the experimental and control group in a training room in Yavuz Selim Family Health Center. Collection of data will take approximately 15-20 minutes. Roma women who are pre-tested will be randomly assigned to the sample pool to be divided into experimental and control groups. Roman women will be divided into experimental and control groups by Simple Random Method.

Data Collection Tools Personal questionnaire; This form was developed in line with the literature and consists of 18 questions to determine the introductory characteristics of the participants. Personal questionnaire includes age, marital status, educational status, income, employment status, social security, family history of cervical cancer, first sexual intercourse age, first birth age, number of births, use of oral contraceptives, gynecological problems, Training status for cervical cancer will be questioned before.

Cervical Cancer and Pap Smear Test Health Belief Model Scale: This scale developed by Champion for breast cancer and mammography; Adapted to Cervical Cancer and Pap Smear Test. The Turkish validity and reliability study was carried out by Güvenç, Akyüz and Açıkel in 2010. The scale consists of 35 items and five main dimensions: sensitivity (3 items), severity (7 items), Pap Smear benefit and motivation (8 items), health motivation (3 items), Pap Smear barriers (14 items). 5-point Likert-type scaling ranging from 1 to 5 in the evaluation of the scale - "strongly disagree" (1), "disagree" (2), "undecided" (3), "agree" (4), "totally agree" (5) - method was used. Each dimension of the scale is evaluated separately and cannot be combined into a single total score. For each individual, points are obtained as much as the number of subscales. The higher the scores, the higher the sensitivity, caring and motivation; It states that the perceived benefits are high for the perception of benefit and the obstacles for the perception of disability are perceived high. Subscales other than the perception of disability subscale are positively associated with Pap Smear screening behavior. The high disability perception score of the individual indicates that the barriers related to having the Pap Smear test are high.

As a result of the research, the data obtained from the personal information form and the cervical cancer and pap smear test health belief model scale will be evaluated in the SPSS package program and will be reported. Descriptive statistics, paired t test, mc nemar test and correlation analysis will be used to evaluate the data. The data recorded with a voice recorder in the focus group meeting will be done by the player. Content analysis will be used in the analysis of the data. Inductive analysis, that is, content analysis based on coding, will be used in content analysis. In this analysis, similar data will be classified under certain concepts and themes and will be interpreted in an understandable way.

Ethical aspects: Study approval was given by Ondokuz Mayıs University Clinical Research Ethics Committee. (Decision No: B.30.2.ODM.0.20.08 / 616-704). All participants were informed about tis study and obtained orat-written informed consents.

ELIGIBILITY:
Inclusion Criteria:

* Being romani
* Be woman
* Being married or living / living with a partner
* To be registered at Yavuz Selim Family Health Center
* 30 years of age or older (to accept as the starting age for scans)
* Being literate
* Not being educated about cervical cancer
* Not having been screened for cervical cancer before
* Not being pregnant or postpartum three-month jobs
* Agree to participate in research
* No communication barriers

Exclusion Criteria:

* Having had problems with the cervix before
* Having a cervical cancer screening
* Having had a hysterectomy operation

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Cervical cancer is one of the cancer types in women.
Enrollment: 80 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Cervical Cancer and Pap Smear Test Health Belief Model Scale: Scale | 3 months
  The scale consists of 35 items and 5 sub-dimensions. Its part of the scale is evaluated separately and cannot be combined into a single total score. Cervical cancer sensitivity sub-dimension consists of 3 items. Hearing score 3-15. The higher the scores, the higher their sensitivity. The benefit and motivation sub-dimension of the Pap smear consists of 8 items. Points 8-40 helpful. An increase in scores indicates an increase in perceptions of benefit and motivation. Cervical cancer health motivation sub-dimension consists of 3 items. Hearing score 3-15. An increase in scores indicates an increased motivation for health. Pap smear barriers sub-dimension consists of 14 items. Scoring 14-70 officer. It means that the higher the scores, the higher the obstacles are perceived. Cervical cancer care / severity sub-dimension consists of 7 items. Hearing score 7-35. Increasing scores indicate an increase in caring / seriousness perceptions.
Focus Group Meeting | 3 months
  A focus group discussion will be held with the participants in the experimental group regarding their educational experiences, learning experiences for cervical cancer and screening, and program outcomes. This evaluation will be completed in 3 sessions, separately for each group.
  Session titles;
  * How did the training and consultancy provided contributed to your learning on the subject?
  * How did the information you get with composed music help you learn the subject?
  * What are the contributions of this training program to your life?
  * How did your experience of music therapy and planned education program affect your awareness of cancer prevention?
  * What and what kind of trainings would you like in future trainings?

CONTACTS AND LOCATIONS:
Overall Officials: İlknur AYDIN AVCİ, Prof, Study Director — Ondokuz Mayıs University
Locations (1):
- Yavuz Selim Family Health Center, Samsun, Turkey (Türkiye)

REFERENCES:
- [Derived] Aydin M, Avci IA. The effect of the music-supported education program on the awareness and health beliefs of Roma women about cervical cancer and screening. BMC Public Health. 2025 Apr 25;25(1):1536. doi: 10.1186/s12889-025-21884-4. PMID 40281521